CLINICAL TRIAL: NCT05145439
Title: A Non-significant Risk Clinical Study to Assess Changes in Perfusion, Oxygenation, and Hemoglobin Content After Application of the VibratoSleeve, a Therapeutic Ultrasound (TUS) Phased Array, for Patients With Ischemic and Neuroischemic Diabetic Foot Ulcers (DFU)
Brief Title: A Non-significant Risk Clinical Study of Therapeutic Ultrasound for Patients With Diabetic Foot Ulcers.
Acronym: Dulcet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vibrato Medical, Inc. (Industry)
Collaborators: Vascular and Interventional Specialists of Orange County, Inc. (VISOC) (Unknown); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S21-003
Record Dates: First submitted 2021-11-10; First posted 2021-12-06 (Actual); Results first posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Foot Ulcer; Peripheral Arterial Disease; Wound; Foot
MeSH Terms: conditions — Diabetic Foot; Peripheral Arterial Disease; Foot Injuries

STUDY DESIGN:
Intervention Model Description: Prospective, single arm, open-label, feasibility acute phase study
Masking Description: Though the treatment device will be known to all participants, the level of treatment will be randomized among 3 distinct sessions and the level of treatment will be masked for the subject (participant), care provider, investigator, and outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- VibratoSleeve TUS (Experimental): In this single arm study, there is only one group/arm, all of whom will be given 3 levels of treatment with the VibratoSleeve TUS device.
  Interventions: Device: VibratoSleeve Therapeutic Ultrasound Device

INTERVENTIONS:
Device: VibratoSleeve Therapeutic Ultrasound Device — The VibratoSleeve is compromised of a 16-transducer array that is mounted within a wrap that conforms to the posterior calf.

SUMMARY:
This study is evaluating whether a therapeutic ultrasound device can improve blood flow to the leg with diabetic foot ulcer (DFU).

DETAILED DESCRIPTION:
The VibratoSleeve TUS will be used on to assess its acute vasodilatory and perfusion effects in diabetic subjects with PAD and DFU. Each subject will receive one 90-minute TUS treatment in each of 3 treatment sessions. All post-treatment acute assessments will take place immediately following each day's treatment and no follow-up assessments will be required in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of at least one DFU (grade 0 or 1 by University of Texas classification)
2. Diagnosis of diabetes mellitus
3. Diagnosis of PAD that meets at least one of the following conditions:

   1. Ankle-brachial index (ABI) of < 0.9 in the same limb as the DFU
   2. Toe Brachial Index (TBI) ≤ 0.6 OR Toe Blood Pressure ≤ 50 mmHg
   3. Documented history of PAD for a minimum of 3 calendar months prior to time of enrollment
4. Aged ≥ 22 years

Exclusion Criteria:

1. Rutherford 6 stage PAD
2. Active DFU infection
3. End-stage renal disease on dialysis
4. HbA1c > 13%.
5. Planned PAD revascularization.
6. Prior stenting in posterior tibial artery.
7. Re-vascularization procedure within 25 days prior to enrollment in the study. (Note: Patients who had re-vascularization procedure earlier than 25 days prior to enrollment are eligible for enrollment if they meet all other criteria).
8. History or diagnosis of severe chronic venous insufficiency or mixed arterio-venous disease.
9. Acute limb ischemia within 30 days prior to treatment.
10. History or diagnosis of deep venous thrombosis below the knee in treatment leg.
11. Any conditions that, in the opinion of the investigator, may render the patient unable to complete the study or lead to difficulties for patient compliance with study requirements, or could confound study data.
12. Patient's enrollment in another investigational study that has not completed the required primary endpoint follow-up period (Note: Patients involved in a long-term surveillance phase of another study are eligible for enrollment in this study).

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-14 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vascular & Interventional Specialists of Orange County, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No
Collective (analyzed) study data will be published with an exception of discussing an individual subject's outcomes (anonymized) that contribute to a better understanding of the treatment.

REFERENCES:
- [Result] Yang C, Weng H, Chen L, Yang H, Luo G, Mai L, Jin G, Yan L. Transcutaneous oxygen pressure measurement in diabetic foot ulcers: mean values and cut-point for wound healing. J Wound Ostomy Continence Nurs. 2013 Nov-Dec;40(6):585-9. doi: 10.1097/WON.0b013e3182a9a7bf. PMID 24202221
- [Result] Kalani M, Brismar K, Fagrell B, Ostergren J, Jorneskog G. Transcutaneous oxygen tension and toe blood pressure as predictors for outcome of diabetic foot ulcers. Diabetes Care. 1999 Jan;22(1):147-51. doi: 10.2337/diacare.22.1.147. PMID 10333917

RESULTS

PARTICIPANT FLOW:
Groups:
- VibratoSleeve TUS: Received treatment with the VibratoSleeve TUS device.
Period: Overall Study
Arm/Group | VibratoSleeve TUS
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | VibratoSleeve TUS
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Transcutaneous oxygen pressure (TcPO2) [Mean (Standard Deviation); unit: mmHg] | 67.54 (17.68)

OUTCOME MEASURES:

1. Primary Outcome: Transcutaneous Oxygen Pressure (TcPO2)
Description: noninvasive test that directly measures the oxygen level of tissue beneath the skin
Time Frame: Through study completion, an average of 1 month.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | VibratoSleeve TUS
Number analyzed (Participants) | 12
mmHg | 50.96 (17.40)

2. Secondary Outcome: Percent Change From Baseline in Perfusion Rate of the Targeted Foot
Description: Calculate percent change in perfusion rate measured non-invasively by Flowmet, compared from baseline to end of treatment.
Time Frame: Through study completion, an average of 1 month
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | VibratoSleeve TUS
Number analyzed (Participants) | 12
Percentage (%) | 34 (4.6)

3. Secondary Outcome: Tissue Oxygen Saturation (StO2)
Description: spatial frequency domain imaging (SFDI) to measure tissue oxygen saturation
Time Frame: Through study completion, an average of 1 month
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | VibratoSleeve TUS
Number analyzed (Participants) | 12
Percentage (%) | 76.0 (17.2)

4. Secondary Outcome: Ankle Brachial Index (ABI)
Description: blood pressure ratio in the upper arm and lower limbs
Time Frame: Through study completion, an average of 1 month
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | VibratoSleeve TUS
Number analyzed (Participants) | 12
ratio | 0.92 (0.026)

ADVERSE EVENTS:
Time Frame: Safety surveillance and reporting starts when subject receives therapy with the VibratoSleeve until the end of the final treatment visit. All treatment visits were completed within an average of 1 month per patient.
Description: Although unlikely due to the nature of the device, the following adverse events were reported for each subject through the final treatment visit:
  * All device-related adverse events and events for which the relationship to the VibratoSleeve is unknown
  * All SAEs Unchanged, chronic, non-worsening or pre-existing conditions are not AEs and should not be reported. Planned hospitalization for a pre-existing condition is not considered a serious adverse event.
Arm/Group | VibratoSleeve TUS
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and Investigator shall have the right to publish data obtained from the Study provided that the Institution and Investigator shall submit copies of any proposed publication or presentation to Sponsor for written approval, for which approval shall not be unreasonably denied. Sponsor reserves the right to delete any Confidential Information or other proprietary information of Sponsor (including trade secrets but not including Results) from the proposed publication or presentation.

DOCUMENTS (1):
  • Study Protocol (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT05145439/Prot_001.pdf